CLINICAL TRIAL: NCT01417949
Title: Immediate Versus Deferred Antiretroviral Therapy in HIV-infected Patients Presenting With Acute AIDS-defining Events (IDEAL-Study)
Brief Title: Immediate Versus Deferred Antiretroviral Therapy in HIV-infected Patients Presenting With Acute AIDS-defining Events
Acronym: IDEAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Nr. 2010-022413-26
Record Dates: First submitted 2011-08-10; First posted 2011-08-16 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-09

CONDITIONS: HIV-Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate arm (Active Comparator): Immediate arm: ART should be initiated as soon as possible but no later than 3 days after initiation of OI treatment.
  Interventions: Other: Time of starting antiretroviral therapy
- Deferred arm (Active Comparator): Deferred arm: ART should be initiated after the completion of OI treatment which is achieved at the earliest at day 21 for PCP and at day 28 for TE. ART should be initiated no later than 6 weeks after initiation of OI treatment.
  Interventions: Other: Time of starting antiretroviral therapy

INTERVENTIONS:
Other: Time of starting antiretroviral therapy — Within 24 hours after sending the screening form, the site investigator will receive a randomization sheet with the decision when to start ART ("immediate" or "deferred"). The day of receiving the randomization sheet will be defined as baseline visit.

SUMMARY:
The purpose of this study is to compare the early versus deferred initiation of antiretroviral combination therapy consisting of tenofovir, emtricitabine and atazanavir/ritonavir in treatment naive patients who present with an acute AIDS-defining illness, namely pneumocystis pneumonia (PCP) or toxoplasma gondii encephalitis (TE).

DETAILED DESCRIPTION:
Objectives:

To compare the early versus deferred initiation of antiretroviral combination therapy consisting of tenofovir, emtricitabine and atazanavir/ritonavir in treatment naive patients who present with an acute AIDS-defining illness, namely pneumocystis pneumonia (PCP) or toxoplasma gondii encephalitis (TE).

The primary objective of this study is as follows:

To compare the rates of clinical progression between both groups. Progression is defined as death, all new/relapsing opportunistic infections (OI), and other grade 4 clinical endpoints (evaluated by standardized toxicity tables) within 24 weeks after randomization.

The secondary objectives of this study are:

* to evaluate and to compare hospitalization days after completion of initial OI treatment between both groups.
* to evaluate the incidence of immune reconstitution inflammatory syndrome (IRIS, definition see Objectives) in both groups during the first 24 weeks.
* to evaluate and to compare the virological outcome proportion in both groups. Virological outcome is assessed by HIV-1 plasma viral load at Week 24 (proportion of patients achieving HIV RNA below 50 copies/mL). For definition of virological failure, see below.
* to evaluate and to compare the frequency changes in ART regimen for lack of efficacy or of toxicity in both groups.
* to evaluate the quality of life (QOL) and the adherence to the ARV regimen in subjects starting tenofovir, emtricitabine and atazanavir/ritonavir at late stages of HIV-1-infection.

Study Design: Prospective, randomized, open-label multicenter study

Number of Subjects to be Randomized:

105 patients per arm (total of 210 patients planned).

Target Population:

ART naïve HIV-1 infected adults, who have developed an acute AIDS defining opportunistic infection, namely PCP or TE.

Duration of Treatment:

24 weeks

Diagnosis and Main Eligibility Criteria:

Key Inclusion Criteria:

* Adult (at least 18 years) HIV-1 infected subjects
* Antiretroviral naïve HIV-1-infected patients who have developed an acute AIDS defining event, namely PCP or TE (women receiving prior MTCT prophylaxis may be enrolled)
* Patients who are able to take or to receive antiretroviral treatment and who are able to give written consent Key exclusion criteria
* Renal failure or CrCl below 60 mL/min
* Patients who are not able to initiate ART or with current contraindications against atazanavir/ritonavir
* Other AIDS-defining events than PCP or TE (exceptions see below)
* Pregnancy/Women of childbearing potential who want to become pregnant

Study Procedures/ Frequency:

OI Diagnosis, Screening, Randomization

* Patients should be screened immediately after diagnosis and decision for OI treatment have been made, providing the patient's personal doctor considers ART to be possible and the patient agrees to be included in the study (written consent).
* Diagnosis of both PCP and TE will be established according to standard of care by the treating physician. A definitive diagnosis (histologically proven) is not required for study entry. The decision for specific treatment of OI is also made by the treating physician according to appropriate guidelines.
* Screening assessments include medical history, social background, physical examination, height, weight, vital signs, and concomitant medications.
* Blood parameters should be assessed by the local lab and should contain CBC (complete blood count) with differential and platelet count, Bilirubine, ALT, AST, LDH, yGT, serum creatinine, electrolytes (sodium, potassium, chloride), calculated creatinine clearance (CrCl), urinalysis, and serum pregnancy test (females of childbearing potential only). These results must be available before sending the evaluation form.
* Further screening assessments include HIV-1 RNA, genotype HIV resistance test, CD4/CD8 T-cell count, serology for hepatitis C antibody, hepatitis B surface antigen (HBsAg), cryptococcus antigen, CRP and a T Cell Interferon-Gamma Release Assay (TIGRA). Of note, there is no need to wait for the results of these further screening parameters.
* A questionnaire that will describe social and educational status and reasons for presenting late during HIV-infection will be performed at screening or entry. A QoL questionnaire (SF 36) is also required at screening or entry.

Randomization, Baseline Prior to first randomization, every participating center will receive study drugs for the treatment of three patients for one month. Within 24 hours after sending the screening form, the site investigator will receive a randomization sheet with the decision when to start ART ("immediate" or "deferred"). The day of receiving the randomization sheet will be defined as baseline visit. Immediate arm: ART should be initiated as soon as possible but no later than 3 days after initiation of OI treatment. Deferred arm: ART should be initiated after the completion of OI treatment which is achieved at the earliest at day 21 for PCP and at day 28 for TE. ART should be initiated no later than 6 weeks after initiation of OI treatment.

Follow up Procedures

* Week 4, 8, 12, 16, 20, 24 or Early Study Drug Discontinuation Visit assessments include a symptom-directed physical examination, weight, vital signs, concomitant medications, adverse events, HIV-1 RNA, CD4 count, CBC with differential and platelet count, ALT, AST, LDH, Bilirubine, gGT, serum creatinine, electrolytes, calculated CrCl.
* Additional Week 12, 24, or Early Study Drug Discontinuation Visit assessments include the preservation of a plasma sample for HIV genotype/phenotype analysis in selected centers. Subjects who were HBsAg positive at screening will have HBV DNA and HBV serology measured at these visits.
* If the subject discontinues study drug prior to Week 24, the subject will be asked to return to the clinic within 72 hours of stopping study drug for an Early Study Drug Discontinuation visit. All of the Week 24 assessments will be performed at this visit.
* HIV resistance assessments will be performed in patients who do not achieve plasma HIV 1 RNA levels of < 400 copies/mL at Week 24, who achieve plasma HIV 1 RNA levels of < 400 copies/mL on at least one occasion, and later have at least two consecutive plasma HIV 1 RNA levels > 400 copies/mL, or for subjects who discontinue study drugs prior to Week 24 and have > 400 copies/mL of HIV 1 RNA on their last study visit prior to discontinuing study drugs.
* Additional Week 12, 24 assessments include a patient adherence questionnaire and a QoL Questionnaire (SF 36).

Test Product, Dose, and Mode of Administration:

Atazanavir capsules with 300 mg and ritonavir tablets with 100 mg, each to be taken QD with a meal. The NRTI backbone chosen by the treating physician is preferably the combination of emtricitabine and tenofovir DF tablets.

Criteria for Evaluation: Primary Endpoint:

Clinical Progression (death, all new or relapsing OI, other Grade 4 clinical endpoint) within 24 weeks. For G4 events standardized toxicity grading tables will be used. For abnormalities not found in the Toxicity Tables, a Grade 4 event will be defined as potentially life-threatening (extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable). Patients who drop out of study observation before end of week 12 are counted as clinical progression.

Secondary Endpoints

* Hospitalization days after completion of OI treatment
* Incidence of immune reconstitution inflammatory syndrome (IRIS) as judged by the site investigator (for definitions see below) compared in the two groups during the first 24 weeks.
* Virological outcome at week 24 (proportion of patients achieving HIV RNA < 400 (<50 copies/mL).
* Proportion of patients with changes in ARV regimen for lack of efficacy or of toxicity
* to evaluate and to compare the immunological outcome proportion in both groups.
* Quality of life (QOL), including overall self-reported QOL at Week 24

Statistical Methods:

Tabular and/or graphical descriptive methods will be used to summarize and explore the results. Continuous variables will be summarized by mean, standard deviation, minimum, 25th, 50th (median), and 75th percentiles and maximum. Count and percent of subjects will summarize categorical variables. Appropriate transformations will be applied (e.g., log10 for HIV-1 RNA). Appropriate confidence intervals (two-sided; 95%) will be calculated for changes in major endpoints. Appropriate tests of significance may also be performed.

This study will be conducted in accordance with the guidelines of Good Clinical Practices (GCPs) including archiving of essential documents.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years) HIV-1 infected subjects
* Antiretroviral naïve HIV-1-infected patients who have developed an acute AIDS defining event, namely PCP or Toxoplasmosis (women receiving prior MTCT prophylaxis may be enrolled)
* Patients who are able to take or to receive antiretroviral treatment and who are able to give written consent

Exclusion Criteria:

* Renal failure or CrCl < 60 mL/min
* Patients who are not able to initiate ART or with current contraindications against atazanavir/ritonavir
* Other AIDS-defining events than PCP or TE (exceptions see below)
* Pregnancy/Women of childbearing potential who want to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Death, all new/relapsing opportunistic infections and other grade 4 clinical endpoints within 24 weeks after randomization | 24 weeks
  Clinical Progression (death, all new or relapsing OI, other Grade 4 clinical endpoint) within 24 weeks. For abnormalities not found in the Toxicity Tables, a Grade 4 event will be defined as potentially life-threatening (extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable). Patients who drop out of study observation before end of week 12 are counted as clinical progression.

SECONDARY OUTCOMES:
Hospitalization days after completion of initial OI treatment between both groups | 24 weeks
  Hospitalization days after completion of OI treatment
incidence of immune reconstitution inflammatory syndrome | 24 weeks
  Incidence of immune reconstitution inflammatory syndrome (IRIS) as judged by the site investigator (for definitions see below) compared in the two groups during the first 24 weeks.
virological outcome | 24 weeks
  Virological outcome at week 24 (proportion of patients achieving HIV RNA < 400 (<50 copies/mL).
efficacy and toxicity of the antiretroviral therapy | 24 weeks
  Proportion of patients with changes in ARV regimen for lack of efficacy or of toxicity
quality of life | 24 weeks
  Quality of life (QOL), including overall self-reported QOL at Week 24
immunological outcome | 24 weeks
  For evaluation of immunological outcome, CD4 T-cell counts at week 24 (absolute, relative, CD4/CD8 ratio) and the change in CD4 T-cell counts from baseline will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schmiedel, MD, Principal Investigator — Infectious Diseases Unit, University Medical Center Hamburg-Eppendorf
Locations (17):
- Germany (17):
  - ICH Study Center GmbH & CO. KG, Hamburg, Hamburg
  - Vivantes Auguste-Viktoria-Klinikum, Berlin, State of Berlin
  - Charitè Universitätsmedizin Berlin Campus Virchow Klinikum, Berlin, State of Berlin
  - Universitätsklinikum Bonn, Innere Medizin I, Immunologische Ambulanz/Studienzentrale, Bonn
  - Universitätsklinik Köln, Klinik I für Innere Medizin, Cologne
  - Medizinische Klinik Nord, Dortmund
  - Universitätsklinikum Düsseldorf, Klinik für Gastroenterologie, Hepatologie und Infektiologie, Düsseldorf
  - Universitätshauptklinik Essen, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik II / Infektiologie, Frankfurt am Main
  - Universitätsklinikum Freiburg, Centrum Chronische Immundefizienz (CCI), Freiburg im Breisgau
  - ifi Hamburg an der Asklepios Klinik St. Georg, Hamburg
  - University Medical Center Hamburg-Eppendorf, Infectious Diseases Unit,, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Immunologie und Rheumatologie, Hanover
  - Universitätsklinikum Kiel, II. Medizinisch Klinik, UKSH, Campus Kiel, Kiel
  - Universitätsklinikum München, Infektionsabteilung, Med. Poliklinik, Klinikum der Universität München, Campus Innenstadt, München
  - Universitätsklinkum Ulm, Comprehensive Infectious Diseases Center (CIDC) Ulm, Sektion Infektiologie und Klinische Immunologie, Zentrum für Innere Medizin, Innere Medizin III, Ulm
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No